CLINICAL TRIAL: NCT02153346
Title: Indirect Cost of Illness Study of Moderate and Severe Asthma in Quebec
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 200347
Record Dates: First submitted 2014-05-22; First posted 2014-06-03 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-06

CONDITIONS: Asthma
Keywords: indirect cost; asthma
MeSH Terms: conditions — Asthma

ARMS (1):
- Arm 1 (Other): Intervention 1 & 2 are associated with Arm 1. All patients enrolled in the study will possibly receive both the valuation of lost productivity and work productivity and activity impairment questionnaires, which are outside of the patient's usual care.
  Interventions: Other: Valuation of lost productivity questionnaire; Other: Work productivity and activity impairment questionnaire

INTERVENTIONS:
Other: Valuation of lost productivity questionnaire — A new, composite questionnaire that can be used to assess the impact of health conditions on lost productivity in monetary units. It measures absenteeism, presenteeism, and non work activities.
Other: Work productivity and activity impairment questionnaire — A six item questionnaire used as a patient-reported quantitative assessment of the amount of absenteeism, presenteeism, and daily activity impairment attributable to a specific health problem.

SUMMARY:
Rationale Asthma is a chronic inflammatory disorder of the airways affecting persons of all ages and is recognized as one of the most common chronic diseases. Canada has one of the highest asthma prevalence rates in the world (8.5%, aged 12 and over) and it is a major cause of hospitalization. The cost of asthma varies dramatically across disease severity, and it is expected that these costs are greater when the condition is sub-optimally managed and controlled. Although a number of publications have been reported on the economic burden of asthma, there is a lack of information on the cost of asthma based on disease severity and level of disease control in Canada. The proposed study aims to i) estimate the annual indirect cost of asthma and ii) the impact of asthma on absenteeism, presenteeism and work productivity in Canada. This information is essential to further quantify the burden of asthma on patients and the healthcare system in the Canadian setting.

Overall Objectives The overall objective of this study is to describe the impact of asthma on patients with moderate to severe asthma and to estimate the indirect costs of asthma care in asthmatic patients followed in tertiary clinics specialized in the field of asthma in Quebec, Canada.

Study Design

A prospective cohort study will be conducted to measure the indirect economical burden of asthma on patients. Patients will be selected and recruited from the BD-Asthma registry and followed prospectively for 1 year. Recruited patients will be asked to complete questionnaires at regular intervals for 1 year to measure indirect cost of disease, using the Valuation of lost productivity (VOLP) questionnaire.

Data Collected For each patient, the following data will be collected

* Patient demographics
* Age
* Sex
* Income
* Level of education
* Smoking
* Disease management and Treatment utilization in the year prior to recruitment
* Physician visits and follow up
* Hospitalizations (number and total days)
* Emergency room visits
* Disease characteristics
* Asthma history
* Year of first diagnosis of asthma severity
* Asthma Control Questionnaire score
* Lung function measures

Data Analysis Methods For each participant, the percentage of time missed from work over a year will be calculated. We will use the human capital approach to calculate the costs of asthma due to lost productivity, incorporating both absenteeism and presenteeism in the calculation of the productivity loss. We will calculate the number of work days in which the person was unable to attend the workplace, and the number of days and percentage of time lost during the days the person's work was affected by their asthma. The fraction of time lost from work in the past year will be multiplied by the average income in Quebec. Finally, this value will be multiplied by the coefficient generated by the VOLP, which reflects the relative value of the productivity loss. In addition, we will calculate the VOLP multiplier for each participant which, combined with the percentage of time missed from work, will create a measure of productivity loss adjusted for the relative importance and replace-ability of the participant's profession.

Sample Size and Power

One hundred subjects will be randomly selected from the BD-Asthma registry.

Limitations

The study population may not be representative of the general asthma population, as moderate to severe asthma will be over represented in these tertiary centers.

DETAILED DESCRIPTION:
Rationale Asthma is a chronic inflammatory disorder of the airways affecting persons of all ages and is recognized as one of the most common chronic diseases. With a continuously increasing prevalence and associated morbidity and mortality, asthma poses a tremendous clinical and economic burden on healthcare systems and on the society as a whole.

According to a report published by the Global Initiative for Asthma (GINA) in 2004 an estimated 300 million people in the world have asthma, and more than 2 million Canadians have asthma. Canada has one of the highest asthma prevalence rates in the world (8.5%, aged 12 and over) and it is a major cause of hospitalization.

The direct and indirect costs associated with asthma are expected to rank among the highest for chronic diseases due to the high prevalence in conjunction with the significant healthcare utilization associated with the disease and the considerable restrictions asthma imposes on the physical, emotional, social, and professional lives of sufferers. The cost of asthma varies dramatically across disease severity, and it is expected that these costs are greater when the condition is sub-optimally managed and controlled. Although a number of publications have been reported on the economic burden of asthma, there is a lack of information on the cost of asthma based on disease severity and level of disease control in Canada. Moreover, no study has compared the annual cost of uncontrolled and "well-controlled" asthma patients. Although population-level direct costs have been previously reported through the use of administrative healthcare databases in various provinces, these databases cannot provide clinical data and are limited to subjects who have a public drug insurance plan.

The proposed study aims to i) estimate the annual indirect cost of asthma and ii) the impact of asthma on absenteeism, presenteeism and work productivity in Canada. This information is essential to further quantify the burden of asthma on patients and the healthcare system in the Canadian setting.

Overall Objectives The overall objective of this study is to describe the impact of asthma on patients with moderate to severe asthma and to estimate the indirect costs of asthma care in asthmatic patients followed in tertiary clinics specialized in the field of asthma in Quebec, Canada.

Primary objectives

* To estimate the annual indirect costs of asthma in asthmatic patients followed in tertiary clinics specialized in the field of asthma in Quebec, Canada
* To estimate the annual indirect cost of asthma by asthma severity and control status (uncontrolled, partly controlled, well controlled) of asthmatic patients followed in tertiary clinics specialized in the field of asthma in Quebec, Canada

Secondary objectives

• To determine the impact of asthma on work productivity in asthmatic patients followed in tertiary clinics specialized in the field of asthma in Quebec, Canada.

Study Design

A prospective cohort study will be conducted to measure the indirect economical burden of asthma on patients. Patients will be selected and recruited from the BD-Asthma registry and followed prospectively for 1 year. Recruited patients will be asked to complete questionnaires at regular intervals for 1 year to measure indirect cost of disease, using the Valuation of lost productivity (VOLP) questionnaire.

Recruitment of patients All eligible patients from the BD-asthma will be invited to participate. Patients approached for participation will be provided verbal and written information on the project and, if the patient agrees to participate, they will be asked to sign the participation consent form. The forms will be collected by the research coordination centre (either at the clinic or the physicians' office or directly with the patient). All recruited eligible patients that have provided their consent will be included in this study.

Source Population The population is defined as individuals diagnosed with asthma (ICD9 codes 493.x).

Study Population The study population is defined as having had at least one diagnosis of asthma (ICD9 codes 493.x) recorded in the BD Asthma database between February 2010 and February 2012.

Clinical information Patient characteristics and clinical information on asthma will be obtained from the BD-asthma database.

Data Collected For each patient, the following data will be collected

* Patient demographics
* Age
* Sex
* Income
* Level of education
* Smoking
* Disease management and Treatment utilization in the year prior to recruitment
* Physician visits and follow up
* Hospitalizations (number and total days)
* Emergency room visits
* Disease characteristics
* Asthma history
* Year of first diagnosis of asthma severity
* Asthma Control Questionnaire score
* Lung function measures

Data Analysis Methods For each participant, the percentage of time missed from work over a year will be calculated. We will use the human capital approach to calculate the costs of asthma due to lost productivity, incorporating both absenteeism and presenteeism in the calculation of the productivity loss. We will calculate the number of work days in which the person was unable to attend the workplace, and the number of days and percentage of time lost during the days the person's work was affected by their asthma. The fraction of time lost from work in the past year will be multiplied by the average income in Quebec. Finally, this value will be multiplied by the coefficient generated by the VOLP, which reflects the relative value of the productivity loss. In addition, we will calculate the VOLP multiplier for each participant which, combined with the percentage of time missed from work, will create a measure of productivity loss adjusted for the relative importance and replace-ability of the participant's profession.

Sample Size and Power

One hundred subjects will be randomly selected from the BD-Asthma registry.

Limitations

The study population may not be representative of the general asthma population, as moderate to severe asthma will be over represented in these tertiary centers.

ELIGIBILITY:
Inclusion Criteria:

* Part of the BD-Asthma registry
* Age 18 years and older
* Patients who signed consent for research with the BD-Asthma registry and signed consent to participate in the indirect cost study.
* Must be alive at the time of recruitment

Exclusion Criteria:

• Patients with a diagnosis of COPD recorded in BD-Asthma at the time of enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-06-22; Primary Completion 2016-04-01 (Actual); Study Completion 2016-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par.) in this cohort study were randomly selected from the BD-Asthma/RESP registry in Quebec, with an asthma diagnosis between June 2014 and January 2015, more than 18 years of age, and followed at the outpatient clinics of Hôpital du Sacré-Coeur de Montréal (HSCM), a tertiary care clinic specialized in asthma.
Pre-assignment Details: 187 participants were selected in the BD-Asthma/RESP database; 160 were contacted of which 101 participants were enrolled in the study. 59 refused to participate. Participants were not assigned to any investigational therapies.
Groups:
- BD-Asthma/RESP: Data was collected by an interview, questionnaires and by review of the medical chart from participants who accepted to be registered in the BD-Asthma/RESP data base.
Period: Overall Study
Arm/Group | BD-Asthma/RESP
Started | 101
Completed | 90
Not Completed | 11
Not completed — Lost to Follow-up | 11

BASELINE CHARACTERISTICS:
Arm/Group | BD-Asthma/RESP
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 36
Education [Number; unit: Participants]
  None | 9
  High school | 27
  College | 15
  University | 41
  missing | 1
Smoking habits [Number; unit: Participants]
  Ex-smokers | 44
  Current smokers | 10
  Never smokers | 46
  missing | 1
Number of years with asthma [Mean (Standard Deviation); unit: Years] | 20.7 (16.7)
Control [Mean (Standard Deviation); unit: ACQ Score] — The Asthma Control Questionnaire (ACQ) is a 7-item questionnaire designed to measure the adequacy of asthma control and the change in asthma control (spontaneous or as a result of treatment). The items score symptoms, FEV1% predicted and daily use of rescue bronchodilator. Each item is scored on a 7 point scale (0=no impairment, 6=maximum impairment). Each item is equally weighted and the total score is the mean of the items (0=totally controlled, 6 severely uncontrolled).
  ACQ Score | 1.4 (0.9)
Age of Asthma onset [Mean (Standard Deviation); unit: Years] | 32.7 (19.1)
FEV1 [Mean (Standard Deviation); unit: Percent predicted] — Within 90 days of registration date
  Percent predicted | 89.3 (23.0)
FEV1/FVC [Mean (Standard Deviation); unit: Percent] — FEV1 is defined as forced expiratory volume in 1 second. FVC is defined as Forced vital capacity.
  Percent | 75.1 (9.4)
BMI [Number; unit: Participants]
  <18.5 | 3
  18.5-24.9 | 18
  25.0-29.9 | 38
  >=30.0 | 39
  missing | 3
Number of years at the HSCM asthma clinic [Mean (Standard Deviation); unit: years] | 10.4 (9.0)
Asthma severity [Number; unit: Participants] — Mild asthma (no asthma medication; low daily dose of ICS monotherapy or LTRA, and Asthma Control Questionnaire (ACQ) < 1.5); Moderate asthma (medium to high daily dose of ICS monotherapy or low to medium daily dose of ICS plus LABA or LTRA, and ACQ < 1.5 or low daily dose ICS monotherapy or LTRA monotherapy, and ACQ ≥ 1.5); Severe asthma (high daily dose of ICS with LABA or LTRAs);Very severe asthma (Omalizumab and/or daily use of prednisone).
  Participants
    Mild | 1
    Moderate | 56
    Severe | 26
    missing | 18
Employment Status [Number; unit: Participants]
  Full time | 37
  Part-time as an employee | 13
  Self-employed | 9
  Work disability | 6
  Unemployed but seeking work | 1
  Retired | 35

OUTCOME MEASURES:

1. Primary Outcome: Indirect Cost of Asthma Per Participant Per 3 Months at Baseline (BL) and 12-month Follow-up (FUP)
Description: Participants completed questionnaires within 2 weeks post-recruitment, 4, 8 and 12 months to measure indirect cost of disease, specifically related to productivity. The following questionnaires were used: WPAI helps to determine presenteeism, absenteeism, and total cost calculation (TCC) possible (number of days during the year of study), while VOLP is used to assess the impact of health conditions on lost productivity in monetary units (United states dollars). The following parameters were calculated: Cost of absenteeism due to asthma (CAA), cost of presenteeism due to asthma (CPA), cost of absenteeism due to asthma in whom TCC was possible (CAA TCC), cost of presenteeism due to asthma in whom TCC was possible (CPA TCC), and total indirect cost due to asthma (TICA).
Time Frame: BL and at 12-month FUP
Population: Source Population: all par. with asthma diagnosed by respirologist and followed at outpatient asthma clinic of the HSCM and registered in BD-Asthma/RESP. Only par. with available data in each category (represented by n=X in the category title) were analyzed. One third of par. selected were retired. Only 59 were active workers (52 at BL; 40 at FUP).
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | BD-Asthma/RESP
Number analyzed (Participants) | 52
US Dollars
  BL, CAA, n=52 | 253.3 (847.5)
  FUP, CAA, n=40 | 70.4 (157.6)
  BL,CPA,n=50 | 16.9 (78.8)
  FUP,CPA, n=39 | 17.1 (37.2)
  BL,CAA TCC, n=46 | 183.3 (648.2)
  FUP,CAA TCC,n=37 | 76.10 (162.64)
  BL,CPA TCC, n=46 | 18.4 (82.0)
  FUP,CPA TCC,n=37 | 17.1 (37.20)
  BL,TICA,n=46 | 201.7 (723.7)
  FUP, TICA, n=37 | 93.2 (182.3)

2. Primary Outcome: Indirect Cost of Asthma by Level of Asthma Control Per Participant Per 3 Months at BL and 12-month FUP
Description: Costs of asthma are greater when the asthma is sub-optimally managed and controlled and varies depending on the par. asthma control. Asthma control was assessed using the Asthma Control Questionnaire (ACQ) and par. were asked to recall their experiences during the previous week and respond to the 6 specified questions on a 7-point Likert scale (0=well-controlled; 6=maximum impairment [poorly controlled]; a score of ≤0.75 indicates well controlled symptoms. The following parameters were presented: Cost of absenteeism due to asthma (CAA), cost of presenteeism due to asthma (CPA), cost of absenteeism due to asthma in whom TCC was possible (CAA TCC), cost of presenteeism due to asthma in whom TCC was possible (CPA TCC), and total indirect cost due to asthma (TICA). Only 59 par. were active workers. When stratified by asthma control and severity each stratum had a sample less than 59. Although results are presented. data may not be reliable due to the low number of par. in each stratum.
Time Frame: BL and 12-month FUP
Population: Source Population. Only participants with available data in each category (represented by n=X in the category title) were analyzed. One third of the participants selected were retired. Only 59 participants were active workers. Therefore the stratification for asthma control and severity included very low numbers (52 at BL; 40 at FUP).
Measure: Mean (Standard Deviation); unit: Canadian Dollars
Groups:
- BD-Asthma/RESP: Data was collected by an interview, questionnaires and by review of the medical chart from participants who accepted to be registered in the BD-Asthma/RESP data base. Only participants actively working who completed the questionnaires were included in the analysis of productivity.
Arm/Group | BD-Asthma/RESP
Number analyzed (Participants) | 52
Canadian Dollars
  BL, Partly controlled, CAA, n=9 | 557.65 (1380.41)
  FUP, Partly controlled, CAA, n=10 | 171.66 (266.70)
  BL, Partly controlled, CPA, n=10 | 57.04 (168.54)
  FUP, Partly controlled, CPA, n=10 | 32.51 (50.72)
  BL, Partly controlled, CAA TCC, n=8 | 585.29 (1473.06)
  FUP, Partly controlled, CAA TCC possible, n=10 | 171.66 (266.70)
  BL,Partly controlled, CPA TCC, n=8 | 71.30 (188.04)
  FUP, Partly controlled, CPA TCC, n=10 | 32.51 (50.72)
  BL, Partly controlled, TICA, n=8 | 656.59 (1660.30)
  FUP, Partly controlled, TICA, n=10 | 204.18 (296.69)
  BL, Uncontrolled, CAA, n=21 | 96.09 (233.01)
  FUP, Uncontrolled, CAA, n=15 | 39.75 (73.72)
  BL, Uncontrolled, CPA, n=22 | 9.20 (34.71)
  FUP, Uncontrolled, CPA, n=14 | 9.34 (25.80)
  BL, Uncontrolled, CAA TCC, n=20 | 100.89 (238.00)
  FUP, Uncontrolled, CAA TCC, n=13 | 45.86 (77.69)
  BL, Uncontrolled, CPA TCC, n=20 | 10.12 (36.36)
  FUP, Uncontrolled, CPA TCC, n=10 | 10.06 (26.71)
  BL, Uncontrolled, TICA, n=20 | 111.01 (239.72)
  FUP, Uncontrolled, TICA, n=13 | 55.92 (99.75)
  BL, Well controlled, CAA, n=22 | 278.92 (949.43)
  FUP, Well controlled, CAA, n=15 | 33.53 (90.66)
  BL,Well controlled, CPA, n=18 | 4.02 (12.84)
  FUP, Well controlled, CPA, n=15 | 11.8 (32.68)
  BL,Well controlled, CAA TCC, n=18 | 96.23 (251.82)
  FUP, Well controlled, CAA TCC, n=14 | 35.92 (93.59)
  BL, Well controlled, CPA TCC, n=18 | 4.02 (12.84)
  FUP, Well controlled, CPA TCC, n=14 | 12.65 (33.74)
  BL,Well controlled, TICA, n=18 | 100.25 (263.14)
  FUP, Well controlled, TICA, n=14 | 48.57 (94.44)

3. Primary Outcome: Indirect Cost of Asthma by Level of Asthma Severity Per Participant Per 3 Months at BL and 12-month FUP
Description: Costs of asthma may vary depending on the participant's asthma severity. Asthma severity was based on the standard definitions for severity and ACQ scores: Mild (<0.75), Moderate (>0.75) and Severe (any ACQ score). The following parameters were presented: Cost of absenteeism due to asthma (CAA), cost of presenteeism due to asthma (CPA), cost of absenteeism due to asthma in whom TCC was possible (CAA TCC), cost of presenteeism due to asthma in whom TCC was possible (CPA TCC), and total indirect cost due to asthma (TICA).
Time Frame: BL and 12-month FUP
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Canadian Dollars
Arm/Group | BD-Asthma/RESP
Number analyzed (Participants) | 52
Canadian Dollars
  BL, Mild, CAA, n=1 | 154.36 (0.00)
  FUP, Mild, CAA, n=1 | 303.74 (0.00)
  BL, Mild, CPA, n=1 | 0.00 (0.00)
  FUP, Mild, CPA n=1 | 0.00 (0.00)
  BL, Mild, CAA TCC, n=1 | 154.36 (0)
  FUP, Mild, CAA TCC, n=1 | 303.74 (0)
  BL, Mild, TICA, n=1 | 154.36 (0.00)
  FUP, Mild, TICA, n=1 | 303.74 (0.00)
  BL, Moderate, CAA, n=30 | 210.09 (803.66)
  FUP, Moderate, CAA, n=21 | 67.75 (160.89)
  BL, Moderate, CPA, n=31 | 8.32 (29.80)
  FUP, Moderate, CPA, n=19 | 8.62 (22.19)
  BL, Moderate, CAA TCC, n=28 | 67.81 (139.95)
  FUP, Moderate, CAA TCC, n=18 | 79.05 (171.85)
  BL, Moderate, CPA TCC, n=28 | 9.21 (31.28)
  FUP, Moderate, CPA TCC, n=18 | 9.10 (22.72)
  BL, Moderate, TICA, n=28 | 77.0 (143.12)
  FUP, Moderate, TICA, n=18 | 88.14 (176.35)
  BL, Severe, CAA, n=10 | 553.96 (1319.40)
  FUP, Severe, CAA, n=7 | 103.16 (229.93)
  BL, Severe, CPA, n=9 | 59.52 (178.57)
  FUP, Severe, CPA, n=8 | 27.99 (54.90)
  BL, Severe, CAA TCC, n=8 | 650.38 (1475.45)
  FUP, Severe, CAA TCC, n=7 | 103.16 (229.93)
  BL, Severe, CPA TCC, n=8 | 66.96 (189.40)
  FUP, Severe, CPA TCC, n=7 | 31.99 (58.03)
  BL, Severe, TICA, n=8 | 717.35 (1661.26)
  FUP, Severe, TICA, n=7 | 135.16 (285.08)

4. Secondary Outcome: Work Productivity Loss as Assessed in Hours Using Work Productivity and Activity Impairment (WPAI) During the Specified Time Points
Description: WPAI is a self-administered instrument to determine the degree to which asthma affected work productivity while at work and affected activities outside of work in the last 7 days and yields 4 types of scores: Absenteeism (work time missed/missed due to other reasons); Presenteeism (actual time worked); Work Productivity Loss (affected productivity while working); and Activity Impairment (affected regular activities). The following parameters were presented: Hours (Hrs) missed due to asthma (HMA), Hrs missed due to other reasons (HMO), and Hrs actually worked (HAW); all in the last 7 days.
Time Frame: At BL, 4-Month, 8-Month and 12-Month FUP
Population: Source Population. Only par. with available data in each category (represented by n=X in the category title) were analyzed. Among the 101 par., 35 (35%) were retired and 59 (58%) were working. Only par. working were who completed the WPAI questionnaire were included in the analysis (56 at BL; 49 at 4 months; 37 at 8 months; 44 at FUP).
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | BD-Asthma/RESP
Number analyzed (Participants) | 56
Hours
  BL, HMA, last 7 days, n=56 | 0.4 (2.8)
  4-Month FUP, HMA, last 7 days, n=49 | 2.4 (9.0)
  8-Month FUP, HMA, last 7 days, n=37 | 0.9 (5.3)
  12-Month FUP, HMA, last 7 days, n=44 | 0.0 (0.3)
  BL, HMO, last 7 days, n=56 | 3.3 (9.0)
  4-Month FUP, HMO, last 7 days, n=49 | 4.2 (9.1)
  8-Month FUP, HMO, last 7 days, n=37 | 6.1 (12.8)
  12-Month FUP, HMO, last 7 days, n=44 | 4.4 (10.5)
  BL, HAW, last 7 days, n=56 | 32.9 (13.4)
  4-Month FUP, HAW, last 7 days, n=49 | 27.6 (15.8)
  8-Month FUP, HAW, last 7 days, n=37 | 28.1 (16.0)
  12-Month FUP, HAW, last 7 days, n=44 | 33.0 (16.6)

ADVERSE EVENTS:
Description: There were no adverse events collected in this study.
Arm/Group | BD-Asthma/RESP
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Important limitations regarding sample size,generalizability and results interpretation.Data not reliable due to low numbers by strata. Changes in work status,full/part-time,and treatments or other factors influencing productivity were not accounted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.